CLINICAL TRIAL: NCT04211038
Title: Assessment of Neural Inspiratory Time Through Transesophageal and Surface Electromyography
Brief Title: Assessment of Neural Inspiratory Time Through sEMG and EMGdi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhenfeng He (Other)
Collaborators: Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Zhenfeng He, principal investigator, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GIRH-201278
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Copd; Ventilation; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy subjects (Experimental): Firstly, increase the inspiratory threshold load step by step(30%-80%MIP),in order to increase neural respiratory drive. Secondly, do incremental cycle ergometry test with the assisstance of NPPV.
  Interventions: Device: inspiratory threshold load device
- COPD subjects (Experimental): Firstly, increase the inspiratory threshold load step by step(30%-80%MIP),in order to increase neural respiratory drive. Secondly, do incremental cycle ergometry test with the assisstance of NPPV.
  Interventions: Device: inspiratory threshold load device

INTERVENTIONS:
Device: inspiratory threshold load device — Before experiment ,every subject use a flanged mouthpiece attached to a manually operated occlusion valve in order to measure maximal inspiratory pressure (MIP)at functional residual capacity .
  And then, the healthy subjects will be increased the neural respiratory drive by increasing the pressure in a water-sealed inspiratory threshold loading device. At last, all subjects will do Incremental cycle ergometry test with the assisstance of NPPV.
  Other Names: cycle ergometer

SUMMARY:
The onset and offset of the neural inspiratory time are fundamentally important measurements in studies of patientventilator interaction, where the level of assistance delivered by the ventilator is controlled by the patient's demand. The onset of neural inspiratory time can be determined in esophageal pressure, transdiaphragmatic pressure, and EMG signals. The investigator compare the onset measured by EMG, esophageal and transdiaphragmatic pressure, and consider that the correlation between them is well in different conditions.

DETAILED DESCRIPTION:
The onset and offset of the neural inspiratory time are fundamentally important measurements in studies of patien-tventilator interaction, where the level of assistance delivered by the ventilator is controlled by the patient's demand. Patient-ventilator asynchrony evaluated using the time lag between onset of the neural inspiratory time and the onset of a mechanical ventilation signal. The onset of neural inspiratory time can be determined in esophageal pressure, transdiaphragmatic pressure, and EMG signals. The investigator compare the onset measured by EMG, esophageal and transdiaphragmatic pressure, and consider that the correlation between them is well in three different conditions.

ELIGIBILITY:
Inclusion Criteria:

* normal cardio-pulmonary function
* without low inspiratory muscle strength
* non-smoker
* without history of the nervous system and respiratory system disease
* sever to very severe stable stage

Exclusion Criteria:

* systemic application of corticosteroids nearly 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-27 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
the onset and duration of neural inspiratory time | through study completion, an average of 5 hours
  Correlation between onsets and duration of measured from espphageal pressure, transdiaphragmatie pressure and EMG.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China